CLINICAL TRIAL: NCT04227041
Title: Single-arm, Prospective, Open-label, Exploratory Study of Pyrotinib Combined With Capecitabine for Metastatic HER-2 Positive Colorectal Cancer Patients After at Least Second-line Standard Treatment
Brief Title: A Study of Pyrotinib Combined With Capecitabine for Metastatic HER-2 Positive Colorectal Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qingdao Zhixin Health Technology Co., Ltd. (Other)
Collaborators: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Principal Investigator, Nailong Yang, Principal Investigator, The Affiliated Hospital of Qingdao University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QingdaoZHT
Record Dates: First submitted 2020-01-10; First posted 2020-01-13 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: HER-2 Positive Colorectal Cancer
MeSH Terms: interventions — pyrotinib; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HER2 positive metastatic colorectal cancer (Experimental)
  Interventions: Drug: Pyrotinib in combination with capecitabine

INTERVENTIONS:
Drug: Pyrotinib in combination with capecitabine — Pyrotinib in combination with capecitabine
  Other Names: Capecitabine

SUMMARY:
To evaluate the efficacy and safety of pyrotinib combined with capecitabine in patients with metastatic her-2 positive colorectal cancer after standard treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients should be histologically diagnosed with metastatic CRC and after receiving at least two standard treatment regimens；
2. Patients with HER2 positive；
3. Metastatic colorectal cancer (stage Ⅳ, T1-4N0-2M1)；
4. Life expectancy is at least 6 months
5. ECOG score 0-1；
6. The functional level of the major organs must meet the following requirements (no blood transfusion within 2 weeks prior to screening, no use of leukocytes or platelets)：

Exclusion Criteria:

1. The histopathological type is mucinous adenocarcinoma or ovarian implant metastasis；
2. Patients who have previously been treated with anti-Her2-targeted drugs；
3. Patients with surgical opportunity or potential for surgical treatment；
4. Patients with a high risk of bleeding or perforation due to a tumor that has apparently invaded adjacent organs (including large vessels) of the colorectal lesion or who have developed fistulas；
5. Patients with any severe and/or uncontrolled disease;
6. Patients with any or present brain metastases；
7. Women who were pregnant or breast-feeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2020-01-10 (Estimated); Primary Completion 2021-01-10 (Estimated); Study Completion 2023-01-10 (Estimated)

PRIMARY OUTCOMES:
Maximally Tolerated Dose (MTD) | up to 36 months
  Evaluation of tumor burden based on RECIST criteria.
Progression-free survival (PFS) | up to 36 months
  Evaluation of tumor burden based on RECIST criteria.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | up to 36 months
  Evaluation of tumor burden based on RECIST criteria.
Duration Of Response (DOR) | up to 36 months
  Evaluation of tumor burden based on RECIST criteria.
Disease Control Rate (DCR) | up to 36 months
  Evaluation of tumor burden based on RECIST criteria.
Incidence of Treatment-Emergent Adverse Events [Safety] | up to 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Qingdao University Hospital, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided